CLINICAL TRIAL: NCT04351204
Title: The MR-Linac Technical Feasibility Protocol For Development of MR-guided Adaptive RadiationTherapy
Brief Title: The MR-Linac Technical Feasibility Protocol
Acronym: UMBRELLA-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Elekta Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N18BREL; NL 65953.031.18 (Registry Identifier: Centrale Commissie Mensgebonden onderzoek)
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Tumors at All Sites Which Will Receive Radiotherapy
Keywords: radiotherapy; MR Linac
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRL (Other): radiotherapy on MR linac
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — multiple new techniques and software for MR-guided adaptive radiation therapy.
  Other Names: MR Linac

SUMMARY:
Radiation therapy is predominantly based on a Computed Tomography (CT) scan obtained during the treatment planning phase. During the course of radiotherapy, however, both the tumor and organs at risk (OAR) are variable in position, shape and size between fractions, and during beam delivery within one treatment fraction. Around the clinical target volume (CTV) a safety margin (Planning Target Volume, PTV) is created to account for these geometric uncertainties to ensure that the tumor receives the prescribed dose.

Direct integration of imaging at the linear accelerator enables daily monitoring of patient positioning, tumor position, and alterations in patient anatomy. Image guided radiotherapy (IGRT) enables the detection and immediate correction of such deviations and increases the precision of delivery.

Adaptive radiotherapy has become an important strategy for serially modifying dose distributions in a manner that can substantially reduce OAR dose and subsequent toxicity, while maintaining adequate target coverage. Current adaptive protocols rely upon a standard CT-based workflow and (cone-beam) CT-based image guidance.

Magnetic Resonance Imaging (MRI) has superior soft-tissue contrast over CT and seems a very promising modality to integrate in the radiation treatment process, facilitating better visualization of the tumor and OAR during treatment.

DETAILED DESCRIPTION:
The proposed protocol aims to determine feasibility of multiple new techniques and software for MR-guided adaptive radiation therapy. For each proposed technique feasibility has to be determined individually. A secondary aim is to prospectively collect data from cohorts of patients treated at the MRL and report on acute toxicity.

By including multiple parallel cohorts, the protocol will accelerate the technical development of MR-guided adaptive radiotherapy and the evidence-based introduction of the MRL into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient, age ≥ 18 years, treated with radiation therapy on the MRL.
* WHO performance 0-2.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Contra-indications for an MRI examination.
* Patient is pregnant.
* Claustrophobia.
* Patients >140 kg and/or a body width > 60 cm.
* Patients with any other clinically significant medical condition which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements or severe psychiatric illness/social situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
technical feasibility | 4 years
  Feasibility of the technical procedure is demonstrated if the technique is successfully applied in 9 out of 10 consecutive patients

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Nowee, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bujold A, Craig T, Jaffray D, Dawson LA. Image-guided radiotherapy: has it influenced patient outcomes? Semin Radiat Oncol. 2012 Jan;22(1):50-61. doi: 10.1016/j.semradonc.2011.09.001. PMID 22177878
- [Result] De Los Santos J, Popple R, Agazaryan N, Bayouth JE, Bissonnette JP, Bucci MK, Dieterich S, Dong L, Forster KM, Indelicato D, Langen K, Lehmann J, Mayr N, Parsai I, Salter W, Tomblyn M, Yuh WT, Chetty IJ. Image guided radiation therapy (IGRT) technologies for radiation therapy localization and delivery. Int J Radiat Oncol Biol Phys. 2013 Sep 1;87(1):33-45. doi: 10.1016/j.ijrobp.2013.02.021. Epub 2013 May 7. No abstract available. PMID 23664076
- [Result] Acharya S, Fischer-Valuck BW, Kashani R, Parikh P, Yang D, Zhao T, Green O, Wooten O, Li HH, Hu Y, Rodriguez V, Olsen L, Robinson C, Michalski J, Mutic S, Olsen J. Online Magnetic Resonance Image Guided Adaptive Radiation Therapy: First Clinical Applications. Int J Radiat Oncol Biol Phys. 2016 Feb 1;94(2):394-403. doi: 10.1016/j.ijrobp.2015.10.015. Epub 2015 Oct 17. PMID 26678659
- [Result] McPartlin AJ, Li XA, Kershaw LE, Heide U, Kerkmeijer L, Lawton C, Mahmood U, Pos F, van As N, van Herk M, Vesprini D, van der Voort van Zyp J, Tree A, Choudhury A; MR-Linac consortium. MRI-guided prostate adaptive radiotherapy - A systematic review. Radiother Oncol. 2016 Jun;119(3):371-80. doi: 10.1016/j.radonc.2016.04.014. Epub 2016 May 6. PMID 27162159
- [Result] Vestergaard A, Hafeez S, Muren LP, Nill S, Hoyer M, Hansen VN, Gronborg C, Pedersen EM, Petersen JB, Huddart R, Oelfke U. The potential of MRI-guided online adaptive re-optimisation in radiotherapy of urinary bladder cancer. Radiother Oncol. 2016 Jan;118(1):154-9. doi: 10.1016/j.radonc.2015.11.003. Epub 2015 Nov 26. PMID 26631646